CLINICAL TRIAL: NCT04382274
Title: Quadratus Lumborum Block Versus Dual Transversus Abdominis Plane and Ilioinguinal/Iliohypogastric Nerve Blocks for Postoperative Analgesia Following Total Abdominal Hysterectomy: A Randomized Controlled Trial
Brief Title: Quadratus Lumborum Block Versus Dual Transversus Abdominis Plane and Ilioinguinal/Iliohypogastric Nerve Blocks for Postoperative Analgesia Following Total Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amr Arafa Elbadry, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: QL versus TAB/II&IH block
Record Dates: First submitted 2020-05-04; First posted 2020-05-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Hysterectomy
Keywords: Hysterectomy; postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadratus Lumborum Block (Experimental): the transducer will be placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border will be visualized, leaving underneath the internal oblique muscle, like a roof over the QL muscle. The probe will be tilted down to identify a bright hyperechoic line that represented the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial then placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle will be proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 20 mL of 0.25% bupivacaine will be applied
  Interventions: Procedure: Quadratus Lumborum Block
- Dual block (Experimental): the probe will be located between the iliac crest and the lower costal margin in the anterior axillary line at the level of umbilicus, and the layers of abdominal wall will be identified (external oblique, internal oblique, and transverse abdominis muscles). In-plane technique will be used and the tip of the needle was inserted between the internal oblique and transverse abdominis muscles. After negative aspiration (to exclude intravascular injection), 20 mL of 0.25% bupivacaine will be injected. Then abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualised between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side.
  Interventions: Procedure: Dual Transversus Abdominis Plane and Ilioinguinal/Iliohypogastric Nerve blocks

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — transducer will be placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border will be visualized leaving underneath the internal oblique muscle, like a roof over the QL muscle. The probe will be tilted down to identify a bright hyperechoic line that represented the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip will be placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle will be proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 20 mL of 0.25% bupivacaine will be applied
  Arms: Quadratus Lumborum Block
Procedure: Dual Transversus Abdominis Plane and Ilioinguinal/Iliohypogastric Nerve blocks — the probe will be located between the iliac crest and the lower costal margin in the anterior axillary line at the level of umbilicus, and the layers of abdominal wall will be identified (external oblique, internal oblique, and transverse abdominis muscles). In-plane technique will be used and the tip of the needle was inserted between the internal oblique and transverse abdominis muscles. After negative aspiration (to exclude intravascular injection), 20 mL of 0.25% bupivacaine will be injected. Then abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualised between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side.
  Arms: Dual block

SUMMARY:
Multimodal pain management program is needed to control severe pain after abdominal hysterectomy which is considered as one of the major abdominal surgeries. Opioids (which are the analgesic of choice) have many adverse effects such as sedation, nausea, and vomiting. Hence, different methods are needed to control pain and decrease opioid consumption and its side effects.

Transversus abdominis plane (TAP) block blocks the sensory afferent nerves run between the abdominal muscles and controls postoperative incisional pain.

Blanco was the first who described the quadratus lumborum block (QLB). Somatic pain after upper and lower abdominal surgery can be controlled by QLB. QLB can be performed for all generations (adult, pediatrics, and pregnant).

QLB is considered to be an easy technique to learn as it is easy to get the key sonoanatomic markers for QLB. The novice can learn this block after only a few performance of the procedure. QLB produces effective postoperative analgesia after abdominal surgery, laparoscopic surgery, anterior abdominal wall surgery, and hip and femur surgery. The analgesic effect of QLB covers 24-48 h. While some authors inserted catheter for continuous infusion of the local anesthetic drug to extend the duration of postoperative analgesia, others added dexamethasone to local anesthetic to extend the effect of local anesthetic drugs.

Ultrasound (US)-guided Ilioinguinal and Iliohypogastric nerve and TAP block have been established as analgesic adjuncts for post hernia repair pain management, under general anaesthesia, neuraxial, MAC and infiltration techniques.

US-guided technique of blocking Ilioinguinal and Iliohypogastric nerves have higher success rate compared to conventional technique. TAP block provides analgesia to the parietal peritoneum and skin of the abdomen in infra-umbilical surgeries. Few cadaveric studies showed good analgesic effect in the region between T10 and L1 following a single posterior TAP injection.

DETAILED DESCRIPTION:
All patients will be assessed preoperatively by history taking, physical examination, and laboratory evaluation. On arrival of the patients to the operative room, electrocardiography, non-invasive blood pressure, pulse oximetry, and capnography will be applied. Baseline parameters such as systolic blood pressure, diastolic blood pressure, mean blood pressure, heart rate (HR), and arterial oxygen saturation will be also recorded.

Intravenous (IV) line will be inserted and IV fluid will be started. For both groups, general anesthesia will be induced with IV injection of fentanyl (1 µg/kg) (Sunny Pharmaceutical, Egypt) and propofol (2mg/kg) (AstraZeneca, UK), and then, atracurium (0.5 mg/kg) (GlaxoSmithKline, UK) will be injected for endotracheal intubation.

Mechanical ventilation will be maintained to keep the end-expiratory CO2 values between 34 and 36 mmHg. Anesthesia will be continued with isoflurane 1%-2% in 100% O2. Incremental dose of atracurium (0.1 mg/kg) will be given every 30 min or when needed.

After endotracheal intubation and before the start of the surgery. A computer system will be used for randomization by creating a list of number each number referred to one of the two groups. Block randomization will be used to ensure equality of the groups. Each number will be sealed in an opaque envelope. Then, each patient will be asked to choose one of the envelopes and give to an anesthesiologist who compared it to the computer-generated list and hence assigned her to one of the two groups. Anesthesiologist (who will be blinded to the collected data until the end of the study) will perform the block techniques and administered the medication.

60 Patients were randomly allocated into two equal groups (each 30 patients):

* Group D-TAP (30 patients): Each patient will receive general anesthesia plus bilateral ultrasound-guided dual TAP [combining TAP and IL/IH nerve blocks]
* Group QL (30 patients): Each patient will receive general anesthesia plus bilateral ultrasound-guided QLB.

Blocks technique:

Both blocks were performed under complete aseptic precautions using ultrasound machine with high-frequency linear probe covered with sterile sheath (Sonoscape® SSI-6000, Chinawith12-6 MHz high-frequency linear probe) and 100-mm needle (B Braun Medical Inc., Bethlehem, PA, USA).

In TAP / Ilioinguinal/Iliohypogastric nerve block, the probe will be located between the iliac crest and the lower costal margin in the anterior axillary line at the level of umbilicus, and the layers of abdominal wall will be identified (external oblique, internal oblique, and transverse abdominis muscles). In-plane technique will be used and the tip of the needle was inserted between the internal oblique and transverse abdominis muscles. After negative aspiration (to exclude intravascular injection), 20 mL of 0.25% bupivacaine will be injected. Then abdomen will be scanned through anterior superior iliac spine (ASIS)-umbilicus line. Ilioinguinal nerve can be visualised between the internal oblique and transverse or external oblique muscles and within 1 to 3 cm from the ASIS. The iliohypogastric nerve lies immediately adjacent. After negative aspiration (to exclude intravascular injection), 10 mL of 0.25% bupivacaine will be injected. The same technique will be performed on the other side.

In QL block, the patient will be positioned supine with lateral tilt to perform the block, and the transducer will be placed at the level of the anterior superior iliac spine and moved cranially until the three abdominal wall muscles will be clearly identified. The external oblique muscle will be followed posterolaterally until its posterior border will be visualized (hook sign), leaving underneath the internal oblique muscle, like a roof over the QL muscle. The probe will be tilted down to identify a bright hyperechoic line that represented the middle layer of the thoracolumbar fascia. The needle will be inserted in plane from anterolateral to posteromedial. The needle tip will be placed between the thoracolumbar fascia and the QL muscle, and after negative aspiration, the correct position of the needle will be proved by injection of 5 mL of normal saline to confirm the space with a hypoechoic image and hydrodissection. An injection of 20 mL of 0.25% bupivacaine will be applied and the same technique will be performed on the other side.

Intraoperative fentanyl 1-2 ug/kg will be given if the HR or the blood pressure or both increase >20% of the baseline. About 30 min before the end of the surgical procedure, paracetamol 1 g IV will be given for all patients. Isoflurane will be discontinued on completion of the surgical procedure, and neostigmine 0.05 mg/kg plus atropine 0.01 mg/kg will be administered to reverse the effect of atracurium. After awakening from anesthesia and achieving an appropriate level of consciousness, the patient will be discharged from the operating room. Visual analog scale (VAS) will be used to assess the postoperative pain; if VAS >3 postoperatively, IV increment of morphine 3 mg will be given. Any side effects were recorded as hypotension (systolic arterial pressure <90 mmHg), arrhythmia, bradycardia (HR <50 beat/min), nausea or vomiting, lower limb muscle weakness, or any other complications.

Measurements:

1. Demographic data as age, BMI, ASA status, duration of anesthesia and duration of surgery
2. Postoperative pain severity assessed by VAS for pain (ranging from 0 to 10, where 0 no pain and 10 maximum pain) will be evaluated postoperatively at 30 min and 2, 4, 6, 12, and 24 h postoperative. Patients with VAS≥ 4 will be received morphine at dose IV increment of morphine 3 mg. while patients with VAS<4 will be received paracetamol 1gm IV infusion.
3. The total dose of morphine used postoperatively/patient (rescue analgesia) within first 24 h postoperative.

   * The total dose of intraoperatively fentanyl.
   * Duration of postoperative analgesia (the time from recovery to the first given dose of morphine)
   * Number of patients needed rescue analgesia.
   * Any recorded postoperative complication as hypotension (systolic arterial pressure <90 mmHg), arrhythmia, bradycardia (HR <50 beat/min), nausea or vomiting, lower limb muscle weakness, or any other complications

ELIGIBILITY:
Inclusion Criteria:

1.60 female patients 2. aged 45-60 years 3. ASA Physical Status Class I and II 4. scheduled for abdominal hysterectomy

Exclusion Criteria:

1. Patients had infection at injection site
2. Allergy to local anesthetics
3. Coagulation disorders
4. Severe obesity
5. Physical or mental diseases which could interfere with the evaluation of pain scores
6. Kidney failure or liver failure.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2020-05-02 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
The total dose of morphine used | up to 24 hours postoperative
  The total dose of morphine used postoperatively/patient (rescue analgesia) within first 24 h postoperative

SECONDARY OUTCOMES:
The total dose of intraoperatively fentanyl | during the procedure/surgery
  The total dose of intraoperatively fentanyl
Duration of postoperative analgesia | up to 24 hours postoperative
  Duration of postoperative analgesia (the time from recovery to the first given dose of morphine)
Number of patients needed rescue analgesia | up to 24 hours postoperative
  Number of patients needed rescue analgesia
Postoperative pain severity | up to 24 hours postoperative
  Postoperative pain severity assessed by Visual Analogue Scale for pain

CONTACTS AND LOCATIONS:
Locations (1):
- Amany Afheem, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No